CLINICAL TRIAL: NCT03834116
Title: The Effect of Resistance Inspiratory Muscle Training in the Management of Breathlessness in Patients With Thoracic Malignancies: A Randomized Controlled Trial
Brief Title: Resistance Inspiratory Muscle Training for Patients With Thoracic Malignancies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: The Affiliated Hospital Of Southwest Medical University (Other)
Responsible Party: Principal Investigator, Professor Alex MOLASIOTIS, Chair Professor of Nursing and Head, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSEARS20180509003
Record Dates: First submitted 2019-02-01; First posted 2019-02-07 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Lung Neoplasm Malignant
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Inspiratory muscle training group (Experimental): A pressure threshold device will be used to deliver IMT, which is commercially available by Phillips Respironics.
  Interventions: Device: Inspiratory muscle training
- Control group (No Intervention): The control group will receive standard treatment in a fast-track design.

INTERVENTIONS:
Device: Inspiratory muscle training — A pressure threshold device will be used to deliver IMT, which is commercially available by Phillips Respironics.
  Arms: Inspiratory muscle training group

SUMMARY:
A small-scale pilot randomized controlled trial conducted by the investigators demonstrated some preliminary evidence that inspiratory muscle training (IMT) could be a promising self-management method for alleviating breathlessness. Hence, the aim of this study is to assess the effectiveness of IMT in patients with thoracic malignancies on dyspnea.

DETAILED DESCRIPTION:
The hypothesis of this study is that inspiratory muscle training (IMT) for a three-month treatment will improve dyspnea in lung cancer patients with stable disease experiencing breathlessness.

Plan of Investigation Subjects The sample will be a heterogeneous group of outpatients cared for in a large university medical center in China (Southwest Medical University Hospital).

Methods The trial will be a two-arm, non-blinded, randomized controlled study. Patients will be randomly assigned through a computer program to IMT or a control group by an independent statistician. The IMT group will receive standard care and additionally the IMT intervention. The control group will receive standard treatment.

Study Design Intervention: A pressure threshold device will be used to deliver IMT, which is commercially available by Phillips Respironics. When patients inhale through the IMT device, the valve blocks air flow until the patient generates sufficient inspiratory pressure to overcome the resistance provided by the spring-loaded valve. The patient must generate the inspiratory pressure, in order for the valve to open and allow inhalation of air. The IMT protocol will have five sessions weekly for 12 weeks for 30 mins/day, divided over two sessions.

Procedures Participants will be recruited at the outpatients' clinic of Southwest Medical University Hospital or referred to the research team by the clinicians. Patients allocated to the experimental arm will have training in the IMT use and the trainer (device) will be adjusted to a level which is comfortable to each patient. In the control arm, patients will be visited for completing the study assessments at the same times as in the experimental arm (months 2 & 3).

Sample Size The investigators have used the mBorg score change [primary outcome] in baseline to month three assessment of 0.80 obtained in the pilot study and the established minimally important difference of 1 for the mBorg to calculate sample size requirements, adding a 25% attrition observed in the pilot study. This corresponds to a sample size of 196 subjects.

Data Processing and Analysis The statistical software package IBM SPSS version 23.0 will be used. Descriptive statistics will summarize the sample characteristics. Generalized estimating equations (GEE) models will be used to compare differential changes in the outcomes between the two study arms across multiple time points (baseline-month 2 and month 3 assessment). A p-value of <0.05 was considered statistically significance. Intention-to-treat analysis will be carried out.

ELIGIBILITY:
Inclusion Criteria:

* adults with histological diagnosis of primary LC or mesothelioma;
* refractory dyspnea not responding to current treatment for the past 2 weeks;
* expected prognosis of >3 months as judged by the clinicians,
* oxygen saturation above 85% at rest.

Exclusion Criteria:

* Those with unstable COPD with frequent or acute exacerbations,
* rapidly worsening dyspnea requiring urgent medical intervention,
* treatment with palliative radiotherapy to the chest received within 4 weeks or chemotherapy within 2 weeks;
* experiencing intractable cough, and those having unstable angina or clinically significant pleural effusion needing drainage

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2019-11-23 (Actual); Primary Completion 2021-09-15 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
Modified Borg Scale (mBorg) | week 8
  It is a vertical 0-10 scale, with corresponding verbal expressions of progressively increased intensity from "nothing at all" to ''maximal."

SECONDARY OUTCOMES:
6-minute walk test (6MWT) | week 8
  6-minute walk test (6MWT) on a level surface, which is easy for patients, well-validated, and correlates well with lung function
6-minute walk test (6MWT) | week 12
  6-minute walk test (6MWT) on a level surface, which is easy for patients, well-validated, and correlates well with lung function
Dyspnea Symptoms and Its Impact on Patients' Functional Status (Dyspnea-12 Questionnaire). | Week 8
  D-12 questionnaire uses 12 items, higher scores indicate more impact of dyspnea on functional status
Dyspnea Symptoms and Its Impact on Patients' Functional Status (Dyspnea-12 Questionnaire). | Week 12
  D-12 questionnaire uses 12 items.
Perceived Severity of Breathlessness | week 8
  Will be measured on a 0-10 numerical rating scale (NRS)
Perceived Severity of Breathlessness | week 12
  Will be measured on a 0-10 numerical rating scale (NRS)
St George's Respiratory Questionnaire | week 8
  The St George's Respiratory Questionnaire will be used. It measures impact on overall health, daily life, and perceived well-being in patients with dyspnea. Scores range from 0 to 100, with higher scores indicating more limitations.
St George's Respiratory Questionnaire | week 12
  The St George's Respiratory Questionnaire will be used. It measures impact on overall health, daily life, and perceived well-being in patients with dyspnea. Scores range from 0 to 100, with higher scores indicating more limitations.
Anxiety and depression | week 8
  The Hospital Anxiety & Depression Scale will be used. It has 14 items, 7 measuring anxiety and 7 measuring depression, with higher scores indicating more anxiety or depression. For each subscale, scores more than 10 indicate clinical signs of anxiety or depression.
Anxiety and depression | week 12
  The Hospital Anxiety & Depression Scale will be used. It has 14 items, 7 measuring anxiety and 7 measuring depression, with higher scores indicating more anxiety or depression. For each subscale, scores more than 10 indicate clinical signs of anxiety or depression.
Modified Borg scale | week 12.
  It is a vertical 0-10 scale, with corresponding verbal expressions of progressively increased intensity from "nothing at all" to ''maximal."
Patients Compliance to IMT Protocol | Week 12.
  Each patient in the experimental arm will be given a training diary to record IMT home practice sessions.

CONTACTS AND LOCATIONS:
Overall Officials: Alex Molassiotis, Study Chair — The Hong Kong Polytechnic University
Locations (1):
- Southwest Medical University Hospital, Luzhou, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barton R, English A, Nabb S, Rigby AS, Johnson MJ. A randomised trial of high vs low intensity training in breathing techniques for breathless patients with malignant lung disease: a feasibility study. Lung Cancer. 2010 Dec;70(3):313-9. doi: 10.1016/j.lungcan.2010.03.007. Epub 2010 Apr 14. PMID 20392515
- [Background] Molassiotis A, Charalambous A, Taylor P, Stamataki Z, Summers Y. The effect of resistance inspiratory muscle training in the management of breathlessness in patients with thoracic malignancies: a feasibility randomised trial. Support Care Cancer. 2015 Jun;23(6):1637-45. doi: 10.1007/s00520-014-2511-x. Epub 2014 Nov 23. PMID 25417042
- [Background] Farquhar MC, Higginson IJ, Fagan P, Booth S. The feasibility of a single-blinded fast-track pragmatic randomised controlled trial of a complex intervention for breathlessness in advanced disease. BMC Palliat Care. 2009 Jul 7;8:9. doi: 10.1186/1472-684X-8-9. PMID 19583857
- [Background] Butland RJ, Pang J, Gross ER, Woodcock AA, Geddes DM. Two-, six-, and 12-minute walking tests in respiratory disease. Br Med J (Clin Res Ed). 1982 May 29;284(6329):1607-8. doi: 10.1136/bmj.284.6329.1607. No abstract available. PMID 6805625
- [Background] Tan JY, Yorke J, Harle A, Smith J, Blackhall F, Pilling M, Molassiotis A. Assessment of Breathlessness in Lung Cancer: Psychometric Properties of the Dyspnea-12 Questionnaire. J Pain Symptom Manage. 2017 Feb;53(2):208-215. doi: 10.1016/j.jpainsymman.2016.08.009. Epub 2016 Oct 5. PMID 27720789
- [Background] Wilcock A, Crosby V, Clarke D, Tattersfield A. Repeatability of breathlessness measurements in cancer patients. Thorax. 1999 Apr;54(4):375. doi: 10.1136/thx.54.4.374b. No abstract available. PMID 10400541
- [Background] Xu W, Collet JP, Shapiro S, Lin Y, Yang T, Wang C, Bourbeau J. Validation and clinical interpretation of the St George's Respiratory Questionnaire among COPD patients, China. Int J Tuberc Lung Dis. 2009 Feb;13(2):181-9. PMID 19146745
- [Background] Walker J, Postma K, McHugh GS, Rush R, Coyle B, Strong V, Sharpe M. Performance of the Hospital Anxiety and Depression Scale as a screening tool for major depressive disorder in cancer patients. J Psychosom Res. 2007 Jul;63(1):83-91. doi: 10.1016/j.jpsychores.2007.01.009. PMID 17586341
- [Derived] Li MY, Liu XL, Peng B, Wang T, Yao LQ, Huang HQ, Kwok WH, Tan JB, Molassiotis A. The effect of resistance inspiratory muscle training in the management of breathlessness in patients with thoracic malignancies: a randomised controlled trial. Support Care Cancer. 2025 May 22;33(6):492. doi: 10.1007/s00520-025-09511-9. PMID 40402333